CLINICAL TRIAL: NCT02285803
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) in Addition to Tinnitus Retraining Therapy (TRT) for Treatment of Chronic Tinnitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZA, Prof., University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 14/40/406
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRT and real tDCS (Active Comparator)
  Interventions: Device: transcranial direct current stimulation (tDCS)
- TRT and sham tDCS (Sham Comparator)
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS)

SUMMARY:
The aim of this study is to evaluate the added effect of tDCS to TRT within patients with chronic, non-pulsatile tinnitus. Patients were randomised in two groups namely, TRT and real tDCS and the second one is TRT with sham tDCS. Evaluations took place at the start of therapy, at the end of the counselling and at last a follow-up visit will be planned after 84 days of the start of the therapy. Subjective outcome measurements such as Tinnitus Functional Index and Visual Analogue Scales of loudness are the primary outcome measurement. Secondary outcome measurements are the Hospital Anxiety and Depression Scale, hyperacusis questionnaire and psychoacoustic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Duration of tinnitus > 6 months
* Maximum loudness of tinnitus on the VAS ≥ 4
* TFI score ≥ 25

Exclusion Criteria:

* Pregnancy
* Psychiatric disorders
* Pace maker or defibrillator
* Pulsatile tinnitus
* Acoustic Neurinoma
* CVA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) | 3 months

SECONDARY OUTCOMES:
Hyperacusis Questionnaire | 3 months
Hospital Anxiety and depression Scale | 3 months
Patient Global Impression of Change | 3 months
Psychoacoustic measurements | 3 months
Late Latency Evoked Potentials | 3 months
Visual Analogue Scale of Loudness | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Rabau S, Van Rompaey V, Van de Heyning P. The effect of Transcranial Direct Current Stimulation in addition to Tinnitus Retraining Therapy for treatment of chronic tinnitus patients: a study protocol for a double-blind controlled randomised trial. Trials. 2015 Nov 10;16:514. doi: 10.1186/s13063-015-1041-2. PMID 26554670